CLINICAL TRIAL: NCT05075941
Title: PREVAC: Evaluation of Vaccination Coverage and Determinants of Success of the COVID-19
Brief Title: Evaluation of Vaccination Coverage and Determinants of Success of the COVID-19 Vaccination Program Among Populations in Very Precarious Situations
Acronym: PREVAC
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Institut de Recherche en Santé Publique, France (Other); Medecins Sans Frontieres, Netherlands (Other); Médecins du Monde (Other); CROIX ROUGE FRANCAISE (Unknown); OBSERVATOIRE DU SAMU SOCIAL (Unknown); INTERLOGEMENT 93 (Unknown); Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-A01960-41
Record Dates: First submitted 2021-10-07; First posted 2021-10-13 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: vaccination coverage; migrants; homeless; travelling community
MeSH Terms: conditions — COVID-19 | interventions — Vaccination Coverage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Shelters Paris/93
  Interventions: Other: Vaccination coverage
- Workers' hostels Paris/93
  Interventions: Other: Vaccination coverage
- travelling community IDF(77/93/95)
  Interventions: Other: Vaccination coverage
- Street/Camps Paris/93
  Interventions: Other: Vaccination coverage
- Covid Homeless and migrants Marseille
  Interventions: Other: Vaccination coverage
- Hostel Paris/93
  Interventions: Other: Vaccination coverage

INTERVENTIONS:
Other: Vaccination coverage — proportion of people declaring to have received at least one dose of vaccination against COVID-19 among target population

SUMMARY:
The main objective of the study is to assess the level of vaccination coverage (VC) against COVID-19 among migrants, homeless and travelling community, according to their living conditions and housing.

The secondary objectives are :

* to compare the estimated level of vaccination coverage in the different sites and strata (emergency shelters/hotels, camps, workers' hostels, on the street) with the estimated level in the general population of the same territory obtained from the French Health Insurance data (SIVAC).
* identify the obstacles and leverage of vaccination (i.e. mobile team) according to living conditions and habitat (socio-demographic factors, personal health history, vaccine adherence, local health policies, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years and older)
* People considered as homeless (homeless, living in a camp or squat) or
* Living in adapted housing (migrant workers' hostel) or
* Housed in residences of the National System or
* Housed in a social residence such as a 115 hotel or a social housing centre
* Freely and voluntarily consenting to participate

Exclusion Criteria:

* Refusal to participate in the study (non-consent).
* Language barrier with no in-person or telephone translation available.
* Impossibility to give free and informed consent (comprehension barrier, cognitive and/or psychiatric and/or addictive disorders, external pressure from family and friends, persons under guardianship, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: migrants, homeless and travelling community
Sampling Method: Non-Probability Sample
Enrollment: 3811 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Vaccination coverage among COVID-19 | one month
  Assess the proportion of people declaring to have received at least one dose of vaccination against COVID-19 among migrants, homeless and travelling community, according to their living conditions and housing
Identify the most appropriate conditions for the use of vaccination against COVID-19 | one month
  Promote interventions to encourage the use of COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth POULET, MD, Principal Investigator — Epicentre
Locations (2):
- France (2):
  - Marseille, Marseille
  - Paris, Paris

IPD SHARING:
Plan to Share IPD: Yes
The results will be presented in a report to the Ministry of Health, the Haute Autorité de Santé and the various partners. The main findings of this study could potentially be compared with the findings of other ongoing studies, once they are completed. An abstract of the findings will be submitted for presentation at a scientific conference, and at least one manuscript will be submitted for publication in a peer-reviewed scientific journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Study partners